CLINICAL TRIAL: NCT02338193
Title: A Randomized Study Evaluating Dapagliflozin and Metformin, Alone and in Combination, in Overweight Women With a Recent History of Gestational Diabetes Mellitus: Effects on Anthropometric Measurements and Cardiometabolic Abnormalities
Brief Title: Dapagliflozin and Metformin,Alone and in Combination, in Overweight/Obese Prior GDM Women
Acronym: DAPA-GDM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Woman's (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Karen Elkind-Hirsch, Director of Research, Woman's
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RP-14-012
Record Dates: First submitted 2015-01-07; First posted 2015-01-14 (Estimated); Results first posted 2019-04-30 (Actual); Last update posted 2019-06-11 (Actual); Status verified 2019-06

CONDITIONS: Diabetes Prevention in Women After GDM Who Are at High-risk
Keywords: GDM; T2DM; prediabetes
MeSH Terms: conditions — Prediabetic State | interventions — dapagliflozin; Metformin

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- DAPA/MET Extended Release (XR) (Experimental): Dapagliflozin plus metformin XR- 5 mg/1000 mg with meal for 4 weeks DAPA/MET XR- 5mg/1000 mg BID final dose for 20 weeks
  Interventions: Drug: DAPA/MET XR
- Dapaglifloxin (Active Comparator): Dapagliflozin- 10 mg once daily before first meal for 24 weeks
  Interventions: Drug: DAPA
- Metformin XR (Active Comparator): Metformin XR with 500 mg once a day for 2 weeks, followed by 500 mg twice a day for 2 weeks, followed by 500 mg in the morning (AM), 1000 mg in the evening ( PM) for 2 weeks, with 1000 mg twice a day as the final dose for 20 weeks
  Interventions: Drug: MET XR

INTERVENTIONS:
Drug: DAPA/MET XR — final dose- 5 mg dapagliflozin/1000 mg glucophage XR BID for 20-24 weeks
  Other Names: Xigduo 5mg/1000 mg
  Arms: DAPA/MET Extended Release (XR)
Drug: DAPA — 10 mg dapagliflozin QD for 20-24 weeks
  Other Names: Farxiga 10 mg
  Arms: Dapaglifloxin
Drug: MET XR — 1000 mg Metformin XR BID for 20-24 weeks
  Other Names: Glucophage XR 500 mg
  Arms: Metformin XR

SUMMARY:
Women with a history of gestational diabetes (GDM) are at substantially increased risk of type 2 diabetes mellitus (T2DM). Compared with the general population, these women are more likely to be overweight or obese. Moreover, weight gain after GDM is significantly associated with T2DM, independent of baseline body weight. Weight gain, particularly increased central adiposity after delivery, is strongly associated with deterioration of β-cell compensation for insulin resistance. Taken together, our findings and other studies support increased abdominal fat as the strongest factor associated with declining B-cell compensation for insulin resistance in prior GDM women at high risk for T2DM. Dapagliflozin is a novel highly selective SGLT2 inhibitor that improves glycemic control by reducing renal glucose reabsorption leading to urinary glucose excretion. Its efficacy and safety has been studied in multiple randomized controlled trials including an add-on to metformin compared with a placebo. To the extent that glucotoxicity contributes to the demise in β-cell function in subjects with impaired glucose, SGLT2 inhibitors also may prove useful in the treatment of "prediabetes." An additional secondary benefit of SGLT2 inhibition is the elimination of calories in the form of glucose. The loss of glucose with attendant caloric loss contributes to weight loss; in addition, improvements in β cell function have been seen. Weight loss seen with SGLT2 inhibitors is similar to that seen with glucagon-like peptide 1 analogs, and may be more acceptable because they are oral agents. A consistent finding in all dapagliflozin studies has been a reduction in blood pressure. The investigators hypothesize that combination dapagliflozin -metformin treatment over a 24-week period will have a greater positive impact on body weight, anthropometric measurements and glycemic and cardiometabolic parameters than dapagliflozin or metformin monotherapy in overweight/obese at-risk women with a history of GDM.

DETAILED DESCRIPTION:
Following written consent, all study patients will undergo the following clinical, metabolic and laboratory evaluations before and during treatment. To ensure that patients remain unidentified, all study subjects will be assigned an individual study identifier which includes the study acronym, patient initials, and unique number. All blood samples will be obtained and results identified and reported using this unique study identifier. A full physical examination will be performed and vital signs (blood pressure, respiration and temperature) determined. Trained personnel using standardized protocols at the baseline and follow-up examination will obtain anthropometric measurements and blood specimens. Absolute body weight, height, waist and hip circumference, body fat distribution (waist/hip {WHR}) and waist/height ratio ({WHtR}) and blood pressure (BP) will be determined. Body weight will be measured to the nearest 0.1 kg using a calibrated digital scale with participants in light clothing and no shoes. Height will be measured to the nearest centimeter. The total body adiposity (total fatness), defined as the accumulation of body fat without regard to regional distribution, will be expressed as BMI and calculated as weight (kg)/ height (m) 2. The circumference measurements will be taken in the upright position using a 15-mm width flexible metric tape held close to the body but not tight enough to indent the skin. Waist circumference (WC) will be measured at the narrowest level midway between the lowest ribs and the iliac crest and hip circumference measured at the widest level over the buttocks while the subjects are standing and breathing normally. The WHR and WHtR will be calculated for measure of body fat distribution.

All patients will randomly be assigned to one of 3 medication treatment groups-- dapagliflozin-metformin (DAP-MET; 5 mg DAP/ MET 1000 mg BID), metformin XR (MET 1000 mg BID) or dapagliflozin (DAP 10 mg QD); all subjects will be allocated to one of these 3 groups based on computer-generated random numbers using a block randomization method. Oral glucose tolerance tests (OGTTs) with glucose (G) and insulin (I) measured at 0, 30, 60, and 120 after glucose load to assess diabetes, fasting (FBG) and mean blood glucose (MBG) concentrations, insulin resistance and pancreatic ß-cell function will be performed prior to randomization and at 20-24 weeks after full doses of study medications are reached. Mean blood glucose (MBG) concentrations will be calculated by summing glucose values obtained at 0,30,60 and 120 minutes during the OGTT and dividing by 4. At the initial lab evaluation, creatinine and calculated eGFR, TSH, and ß-hCG will be determined for study inclusion. Baseline blood samples will also be analyzed for lipid profiles and liver enzymes.

All patients will receive the same counseling concerning the benefits of lifestyle modification through diet and exercise. The patients will be also encouraged to increase daily exercise (such as walking, using stairs), although this will not be formally assessed. The participants will receive further encouragement to adhere to the regime during follow-up phone calls. Side effects of the treatment and reason for any withdrawals from the study will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* • Overweight/obese (BMI >25) females 18 years to 45 years of age, who experienced gestational diabetes (GDM) during recent (within 12 months) pregnancy

  * postpartum metabolic abnormalities determined by a 75 g oral glucose tolerance test (Inclusive of prior GDM women with impaired fasting glucose (IFG), impaired glucose tolerance (IGT), or both (IFG/IGT) postpartum)
  * Completed lactation
  * Using adequate contraception during study period unless sterilized
  * Written consent for participation in the study

Exclusion Criteria:

* Cholestasis during the past pregnancy
* Any hepatic diseases in the past (viral hepatitis, toxic hepatic damage, jaundice of unknown etiology), gallstones, abnormal liver function tests or renal impairment (elevated serum creatinine levels or abnormal creatinine clearance
* Presence of significant systemic disease, heart problems including congestive heart failure, history of pancreatitis, or diabetes mellitus (Type 1 or 2)
* Renal impairment (e.g., serum creatinine levels ≥1.4 mg/dL for women, or eGFR <60)
* Significantly elevated triglyceride levels (fasting triglyceride > 400 mg %)
* Untreated or poorly controlled hypertension (sitting blood pressure >160/95mm Hg)
* Prior history of a malignant disease requiring chemotherapy
* Known hypersensitivity or contraindications to use of insulin sensitizers such as metformin or thiazolidinediones
* History of hypersensitivity reaction to dapagliflozin or other SGLT2 inhibitors (e.g. anaphylaxis, angioedema, exfoliative skin conditions)
* Current use of metformin, thiazolidinediones, GLP-1 receptor agonists, DPP-4 inhibitors, SGLT2 inhibitors or weight loss medications (prescription or OTC)
* Uncontrolled thyroid disease (documented normal TSH) or hyperprolactinemia
* Liver enzymes (serum alanine aminotransferase [ALT] and/or aspartate aminotransferase [AST] ) levels exceeding more than twice normal lab values
* Use of drugs known to exacerbate glucose tolerance
* History of diabetes or prior use of medications to treat diabetes except GDM
* Currently lactating
* Eating disorders (anorexia, bulimia) or gastrointestinal disorders
* Suspected pregnancy (documented negative serum pregnancy test within 72 hours before first dose of study drug), desiring pregnancy in next 6 months, breastfeeding, or known pregnancy in last 2 months
* Active or prior history of substance abuse (smoke or tobacco use within past 3 years) or significant intake of alcohol or history of alcoholism
* Patient not willing to use adequate contraception during study period and up to 4 weeks after last dose of study drug (unless sterilized).
* Debilitating psychiatric disorder such as psychosis or neurological condition that might confound outcome variables
* Inability or refusal to comply with protocol
* Not currently participating or having participated in an experimental drug study in previous three months

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 69 (Actual)
Dates: Start 2015-09-22 (Actual); Primary Completion 2019-02-13 (Actual); Study Completion 2019-03-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen E Elkind-Hirsch, PhD, Principal Investigator — Woman's Hospital, Louisiana; Renee Harris, MD, Principal Investigator — Woman's Hospital, Louisiana
Locations (1):
- Woman's Hospital, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No
Will publish findings. Individual patient information will be revealed only to patient

REFERENCES:
- [Derived] Elkind-Hirsch KE, Seidemann E, Harris R. A randomized trial of dapagliflozin and metformin, alone and combined, in overweight women after gestational diabetes mellitus. Am J Obstet Gynecol MFM. 2020 Aug;2(3):100139. doi: 10.1016/j.ajogmf.2020.100139. Epub 2020 May 16. PMID 33345876

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients recruited from Woman's Hospital post delivery
Pre-assignment Details: 3 patients not randomized since reluctant to take medication
Groups:
- DAPA/MET XR: Dapagliflozin plus metformin XR- 5 mg/1000 mg with meal for 4 weeks DAPA/MET XR- 5mg/1000 mg BID final dose for 20 weeks
  DAPA/MET XR: final dose- 5 mg dapagliflozin/1000 mg glucophage XR BID for 20-24 weeks
- Metformin XR: Metformin XR with 500 mg once a day for 2 weeks, followed by 500 mg twice a day for 2 weeks, followed by 500 mg in the AM, 1000 mg in the PM for 2 weeks, with 1000 mg twice a day as the final dose for 20 weeks
  MET XR: 1000 mg Metformin XR BID for 20-24 weeks
Period: Overall Study
Arm/Group | DAPA/MET XR | Dapaglifloxin | Metformin XR
Started | 20 | 21 | 25
Completed | 17 | 17 | 15
Not Completed | 3 | 4 | 10
Not completed — Withdrawal by Subject | 0 | 0 | 2
Not completed — Pregnancy | 0 | 1 | 1
Not completed — Noncompliant with visits | 2 | 2 | 7
Not completed — moved out of state | 0 | 1 | 0
Not completed — intolerant of side effects | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: within 1 year postpartum of GDM pregnancy
Groups:
- Total: Total of all reporting groups
Arm/Group | DAPA/MET XR | Dapaglifloxin | Metformin XR | Total
Number analyzed (Participants) | 20 | 21 | 25 | 66
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 20 | 21 | 25 | 66
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 21 | 25 | 66
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 20 | 21 | 25 | 66
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 6 | 6 | 10 | 22
  White | 14 | 15 | 15 | 44
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 21 | 25 | 66
BMI greater than/equal to 25 [Count of Participants; unit: Participants] | 20 | 21 | 25 | 66

OUTCOME MEASURES:

1. Primary Outcome: Change in Body Weight
Description: Change in absolute body weight with combination therapy compared to monotherapy from baseline to week 24
Time Frame: Change from baseline (time 0) to study end (24 weeks)
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | DAPA/MET XR | Dapaglifloxin | Metformin XR
Number analyzed (Participants) | 17 | 17 | 15
kilograms | -21.5 (14) | -12.5 (20) | -4.4 (18)
Statistical Analysis 1: Comparison: DAPA/MET XR vs Dapaglifloxin vs Metformin XR; One Way ANOVA with Bonferroni contrast if p>0.05; Test type: Superiority; p < 0.032, ANOVA

2. Secondary Outcome: Change in Percent Body Weight
Description: Change in percent body weight with combination therapy compared to monotherapy from baseline to week 24
Time Frame: Change from baseline (time 0) to study end (24 weeks)
Measure: Mean (Standard Deviation); unit: percent weight loss from baseline
Arm/Group | DAPA/MET XR | Dapaglifloxin | Metformin XR
Number analyzed (Participants) | 17 | 17 | 15
percent weight loss from baseline | -4.9 (3.1) | -3.2 (4.5) | -1.1 (4.4)
Statistical Analysis 1: Comparison: DAPA/MET XR vs Metformin XR; Test type: Superiority; p < 0.05, ANOVA; One Way ANOVA with Bonferoni contrast test

3. Secondary Outcome: Body Mass Index (BMI)
Description: BMI (measure of overall adiposity) in combination therapy compared to monotherapy after 24 weeks of treatment
Time Frame: 24 weeks of treatment
Measure: Mean (Standard Deviation); unit: kg/m2
Arm/Group | DAPA/MET XR | Dapaglifloxin | Metformin XR
Number analyzed (Participants) | 17 | 17 | 15
kg/m2 | 33 (6.2) | 33.7 (7.7) | 31 (5.4)
Statistical Analysis 1: Comparison: DAPA/MET XR vs Dapaglifloxin vs Metformin XR; Factorial repeated measures ANOVA with Bonferroni contrast test; Test type: Superiority; p < 0.01, ANOVA

4. Secondary Outcome: Waist Circumference (WC)
Description: Waist size (measure of truncal adiposity)with combination therapy compared to monotherapy after 24 weeks of treatment
Time Frame: 24 weeks of treatment
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | DAPA/MET XR | Dapaglifloxin | Metformin XR
Number analyzed (Participants) | 17 | 17 | 15
centimeters | 95.6 (12.7) | 95 (16.6) | 91.7 (11.4)
Statistical Analysis 1: Comparison: DAPA/MET XR vs Dapaglifloxin vs Metformin XR; Factorial repeated measures ANOVA with Bonferroni contrast test; Test type: Superiority; p < 0.012, ANOVA

5. Secondary Outcome: Waist- to -Hip Ratio (WHR; Measure of Central Adiposity)
Description: Waist-to-hip ratio with combination therapy compared to monotherapy after 24 weeks of treatment
Time Frame: 24 weeks of treatment
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | DAPA/MET XR | Dapaglifloxin | Metformin XR
Number analyzed (Participants) | 17 | 17 | 15
Ratio | 0.81 (0.055) | 0.80 (.06) | 0.83 (.06)
Statistical Analysis 1: Comparison: DAPA/MET XR vs Dapaglifloxin vs Metformin XR; Factorial repeated measures ANOVA with Bonferroni contrast test; Test type: Superiority; p = 0.007, ANOVA

6. Secondary Outcome: Waist-to-height Ratio (WHtR)
Description: Waist divided by height a( measure of central adiposity) with combination therapy compared to monotherapy after 24 weeks of therapy
Time Frame: 24 weeks of treatment
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | DAPA/MET XR | Dapaglifloxin | Metformin XR
Number analyzed (Participants) | 17 | 17 | 15
ratio | 0.58 (.06) | 0.57 (.09) | 0.56 (.06)
Statistical Analysis 1: Comparison: DAPA/MET XR vs Dapaglifloxin vs Metformin XR; Factorial repeated measures ANOVA with Bonferroni contrast; Test type: Superiority; p = 0.023, ANOVA

7. Secondary Outcome: Diastolic Blood Pressure (DBP)
Description: Diastolic blood pressure with combination therapy compared to monotherapy after 24 weeks of treatment
Time Frame: 24 weeks of treatment)
Measure: Mean (Standard Deviation); unit: mmHG
Arm/Group | DAPA/MET XR | Dapaglifloxin | Metformin XR
Number analyzed (Participants) | 17 | 17 | 15
mmHG | 79 (11) | 77.8 (11) | 79 (7.5)
Statistical Analysis 1: Comparison: DAPA/MET XR vs Dapaglifloxin vs Metformin XR; Factorial repeated measures ANOVA with Bonferroni contrast; Test type: Superiority; p > 0.05, ANOVA

8. Secondary Outcome: Systolic Blood Pressure (SBP)
Description: Systolic blood pressure with combination therapy compared to monotherapy after 24 weeks of therapy
Time Frame: 24 weeks of treatment
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | DAPA/MET XR | Dapaglifloxin | Metformin XR
Number analyzed (Participants) | 17 | 17 | 15
mmHg | 125 (12) | 124 (13) | 119.6 (10.4)
Statistical Analysis 1: Comparison: DAPA/MET XR vs Dapaglifloxin vs Metformin XR; Factorial repeated measures ANOVA with Bonferroni contrast; Test type: Superiority; p > 0.05, ANOVA

9. Secondary Outcome: Liver Enzymes
Description: ALT/AST ratio with combination therapy compared to monotherapy after 24 weeks of treatment
Time Frame: 24 weeks of treatment
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | DAPA/MET XR | Dapaglifloxin | Metformin XR
Number analyzed (Participants) | 17 | 17 | 15
Ratio | 1.13 (.35) | 1.12 (.32) | 1.18 (.3)
Statistical Analysis 1: Comparison: DAPA/MET XR vs Dapaglifloxin vs Metformin XR; Factorial repeated measures ANOVA with Bonferroni contrast; Test type: Superiority; p < 0.001, ANOVA

10. Secondary Outcome: Total Cholesterol Levels (CHOL)
Description: Cholesterol levels with combination therapy compared to monotherapy after 24 weeks of treatment
Time Frame: 24 weeks of treatment
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | DAPA/MET XR | Dapaglifloxin | Metformin XR
Number analyzed (Participants) | 17 | 17 | 15
mg/dL | 196 (45) | 168 (32) | 178 (31)
Statistical Analysis 1: Comparison: DAPA/MET XR vs Dapaglifloxin vs Metformin XR; Factorial repeated measures ANOVA with Bonferroni contrast test; Test type: Superiority; p < 0.001, ANOVA

11. Secondary Outcome: Triglyceride (TRG) Levels
Description: Triglyceride levels with combination therapy compared to monotherapy after 24 weeks of treatment
Time Frame: 24 weeks of treatment
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | DAPA/MET XR | Dapaglifloxin | Metformin XR
Number analyzed (Participants) | 17 | 17 | 15
mg/dL | 119 (59) | 89.8 (39) | 212 (64)
Statistical Analysis 1: Comparison: DAPA/MET XR vs Dapaglifloxin vs Metformin XR; Factorial repeated measures ANOVA with Bonferroni contrast test; Test type: Superiority; p < 0.004, ANOVA

12. Secondary Outcome: Fasting Blood Glucose (FBG)
Description: Fasting blood glucose levels with combination therapy compared to monotherapy after 24 weeks of treatment
Time Frame: 24 weeks of treatment
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | DAPA/MET XR | Dapaglifloxin | Metformin XR
Number analyzed (Participants) | 17 | 17 | 15
mg/dL | 89 (7.9) | 91 (9.2) | 87 (4.3)
Statistical Analysis 1: Comparison: DAPA/MET XR vs Dapaglifloxin vs Metformin XR; Factorial repeated measures ANOVA with Bonferroni contrast test; Test type: Superiority; p < 0.02, ANOVA

13. Secondary Outcome: Mean Blood Glucose (MBG) During an OGTT
Description: Mean blood glucose after glucose load with combination therapy compared to monotherapy after 24 weeks of treatment
Time Frame: 24 weeks of treatment
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | DAPA/MET XR | Dapaglifloxin | Metformin XR
Number analyzed (Participants) | 17 | 17 | 15
mg/dL | 109.5 (15.2) | 110.1 (17.8) | 112.5 (15)
Statistical Analysis 1: Comparison: DAPA/MET XR vs Dapaglifloxin vs Metformin XR; Factorial repeated measures ANOVA with Bonferroni contrast test; Test type: Superiority; p < 0.012, ANOVA

14. Secondary Outcome: Fasting Insulin Sensitivity (HOMA-IR)
Description: HOMA index of insulin resistance calculated from fasting insulin and glucose with combination therapy compared to monotherapy after 24 weeks of treatment
Time Frame: 24 weeks of treatment
Measure: Mean (Standard Deviation); unit: Index
Arm/Group | DAPA/MET XR | Dapaglifloxin | Metformin XR
Number analyzed (Participants) | 17 | 17 | 15
Index | 2.6 (1.6) | 2.4 (1.4) | 1.8 (0.84)
Statistical Analysis 1: Comparison: DAPA/MET XR vs Dapaglifloxin vs Metformin XR; Factorial repeated measures ANOVA with Bonferroni contrast test; Test type: Superiority; p > 0.05, ANOVA

15. Secondary Outcome: Matsuda Sensitivity Index (SI OGTT)
Description: Surrogate measure of insulin sensitivity derived from OGTT with combination therapy compared to monotherapy after 24 weeks of treatment
Time Frame: 24 weeks of treatment
Measure: Mean (Standard Deviation); unit: Index
Arm/Group | DAPA/MET XR | Dapaglifloxin | Metformin XR
Number analyzed (Participants) | 17 | 17 | 15
Index | 6.0 (3.2) | 6.3 (4.4) | 5.42 (2.4)
Statistical Analysis 1: Comparison: DAPA/MET XR vs Dapaglifloxin vs Metformin XR; Factorial repeated measures ANOVA with Bonferroni contrast test; Test type: Superiority; p < 0.028, ANOVA

16. Secondary Outcome: First Phase Insulin Secretion (IGI/HOMA-IR)
Description: Corrected early insulin response to glucose challenge [(insulinogenic index (IGI)/ divided by fasting insulin resistance index (HOMA-IR)] with combination therapy compared to monotherapy after 24 weeks of treatment
Time Frame: 24 weeks of treatment
Measure: Mean (Standard Deviation); unit: Index
Arm/Group | DAPA/MET XR | Dapaglifloxin | Metformin XR
Number analyzed (Participants) | 17 | 17 | 15
Index | 1.7 (3.2) | 1.1 (1.2) | 0.77 (.53)
Statistical Analysis 1: Comparison: DAPA/MET XR vs Dapaglifloxin vs Metformin XR; Factorial repeated measures ANOVA with Bonferroni contrast test; Test type: Superiority; p < .03, ANOVA

ADVERSE EVENTS:
Time Frame: 6 months while participating in trial
Arm/Group | DAPA/MET XR | Dapaglifloxin | Metformin XR
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/21 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/21 | 0/25
Other Adverse Events (participants affected / at risk) | 6/20 | 6/21 | 5/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DAPA/MET XR (N=20) | Dapaglifloxin (N=21) | Metformin XR (N=25)
Yeast infection (Renal and urinary disorders) | 5 (5) | 6 (6) | 0 (0)
Nausea/diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 5 (5)

LIMITATIONS AND CAVEATS:
Important limitations were the small number completed patients per drug group and only 24 weeks of therapy. Surrogate measures were for central adiposity; use of dual-energy x-ray absorptiometry to measure body composition would increase accuracy

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2018-08-31): https://cdn.clinicaltrials.gov/large-docs/93/NCT02338193/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2018-07-10): https://cdn.clinicaltrials.gov/large-docs/93/NCT02338193/Prot_SAP_001.pdf